CLINICAL TRIAL: NCT00000670
Title: Safety and Tolerance of Zidovudine With Probenecid and the Effect of Probenecid on Zidovudine Pharmacokinetics Over Four Weeks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 107; 11082 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Probenecid; Drug Evaluation; Drug Interactions; Acquired Immunodeficiency Syndrome; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Probenecid; Zidovudine

INTERVENTIONS:
Drug: Probenecid
Drug: Zidovudine

SUMMARY:
To evaluate the interaction of probenecid with zidovudine (AZT). Because AZT is eliminated quickly from the body, it must be taken frequently. A previous study showed that probenecid slowed the elimination of AZT without side effects, but that study lasted only 5 days. This study is to see whether this effect continues for 1 month and whether the continuation of probenecid and AZT is free of side effects over 1 month.

DETAILED DESCRIPTION:
Because AZT is eliminated quickly from the body, it must be taken frequently. A previous study showed that probenecid slowed the elimination of AZT without side effects, but that study lasted only 5 days. This study is to see whether this effect continues for 1 month and whether the continuation of probenecid and AZT is free of side effects over 1 month.

Patients are hospitalized overnight on three separate occasions. On the first admission, AZT is administered every 4 hours. On the second day, 15 blood samples are taken to determine how fast the AZT enters and is removed from the bloodstream (pharmacokinetics). On the second day, after all the blood specimens have been collected, patient starts taking probenecid by mouth every 8 hours, and is discharged from the research unit. The AZT dose is then taken every 8 hours. One week later and again 3 weeks after that, patient is readmitted overnight and the blood sampling to measure AZT levels is repeated. AMENDED: 8 additional patients will be enrolled using the same doses of AZT but a lower dose of probenecid.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Interferon.
* Aerosolized pentamidine for Pneumocystis carinii pneumonia (PCP) prophylaxis.

Concurrent Treatment:

Allowed:

* Radiation for skin lesions.

Patients with symptomatic HIV infection taking zidovudine (AZT) five or six times a day as therapy. Includes patients with AIDS who have history of cytologically confirmed Pneumocystis carinii pneumonia (PCP), patients with advanced AIDS related complex (ARC), and HIV antibody positive patients.

Patients must be able to give written informed consent.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Allergy to probenecid.
* Any underlying medical condition sufficient, in the investigator's opinion, to prevent adequate compliance with study therapy.
* History of urinary tract urate stones or gout.
* Becoming acutely ill, unstable, or febrile.

Concurrent Medication:

Excluded:

* Methotrexate.
* Antiretroviral drugs.
* Ganciclovir.
* Amphotericin.
* Experimental drugs.
* Isoniazid.
* Pyrazinamide.
* Flucytosine.
* Intravenous pentamidine.
* Dapsone.
* Fansidar.
* Antineoplastic drugs not specifically allowed.
* Trimethoprim / sulfamethoxazole.
* Valproic acid.
* Opiates.
* Rifampin.
* Sulfonylureas.

Concurrent Treatment:

Excluded:

* Radiation not specifically allowed.

Patients with the following are excluded:

* Allergy to probenecid.
* Any underlying medical condition sufficient, in investigator's opinion, to prevent adequate compliance with study therapy.
* History of urinary tract urate stones or gout.
* Becoming acutely ill, unstable, or febrile.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16
Dates: Study Completion 1989-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: BG Petty, Study Chair; DM Kornhauser, Study Chair; PS Lietman, Study Chair; JG Bartlett, Study Chair
Locations (2):
- United States (2):
  - UCD Med Ctr, Sacramento, California
  - Johns Hopkins Hosp, Baltimore, Maryland

REFERENCES:
- [Background] Wong SL, Hedaya MA, Sawchuk RJ. Competitive inhibition of zidovudine clearance by probenecid during continuous coadministration. Pharm Res. 1992 Feb;9(2):228-35. doi: 10.1023/a:1018993524818. PMID 1553347